CLINICAL TRIAL: NCT02357277
Title: The Effects of Inhaled Glucocorticoids on the Postmenopausal Skeleton
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAO5309
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Glucocorticoids; Postmenopausal
MeSH Terms: conditions — Osteoporosis | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Budesonide 360 mcg (Experimental): Budesonide dry powder inhaler 2 puffs of 90 mcg twice daily for 4 weeks
  Interventions: Drug: Budesonide
- Budesonide 720 mcg (Experimental): Budesonide dry powder inhaler 2 puffs of 180 mcg twice daily for 4 weeks
  Interventions: Drug: Budesonide
- Placebo (Placebo Comparator): Placebo inhaler 2 puffs twice daily for 4 weeks
  Interventions: Other: Placebo Inhaler

INTERVENTIONS:
Drug: Budesonide — inhaled glucocorticoid budesonide as dry powder inhaler
  Other Names: Pulmicort flexhaler
  Arms: Budesonide 360 mcg; Budesonide 720 mcg
Other: Placebo Inhaler — inhaled placebo
  Arms: Placebo

SUMMARY:
There are over 10 million individuals with asthma using inhaled glucocorticoids (IGCs) in the United States. While oral GCs are recognized to have destructive skeletal effects, far less is known about the effects of IGCs. This gap in our knowledge is of critical importance, not only because of the prevalence, chronic nature and long duration of IGC use, but also because several studies have found that patients using IGCs are at increased risk of fracture. Fracture risk is greatest in postmenopausal (PM) women, in whom IGCs may augment negative effects of estrogen loss and aging.

The investigators hypothesize that initiation of IGCs in IGC naïve PM women will lead to decreased bone formation and uncoupling of bone turnover, a potential mechanism for the effect of IGCs on the skeleton.

To test our hypothesis, the investigators will perform a randomized, controlled 4 week study of the acute effects of commonly used doses of budesonide (360 or 720 mcg) on bone turnover and circulating osteoblast precursors in 60 treatment naïve, non-asthmatic, PM women. These studies are of high clinical significance because there are currently no guidelines regarding screening, prevention or treatment for osteoporosis in patients using IGCs, nor is IGC use taken into account when calculating fracture risk in PM women, the group at highest risk of fracture. High quality evidence for low volumetric bone mineral density (BMD) and abnormal bone quality in PM women using IGCs has the potential to change clinical practice by supporting specific interventions to prevent bone loss and fractures.

DETAILED DESCRIPTION:
The investigators will study acute biochemical and hormonal responses over 4 weeks to commonly prescribed moderate and high doses of budesonide one of the most widely prescribed IGCs, and the preferred drug for Medicare and Medicaid. Sixty treatment naïve PM non-asthmatic women will be randomized to one of 3 groups (20/group): placebo, budesonide 360 or 720 mcg/day. IGCs will be self-administered as 2 puffs twice daily. Budesonide will be provided as Pulmicort flexhaler. At the baseline visit, subjects will be taught proper technique for self-administration of the inhaled medications, including mouth rinsing after each dose. Since dry powder formulations will be used, spacer devices are not required. Women will be assessed at baseline, 1,2, and 4 weeks. This time period and schedule was chosen to ensure adequate time for IGCs to reach peak levels, and to assess the bone metabolic response. Given the 4-6 hr half-life of budesonide, steady state pharmacokinetics will be reached at one week. The investigators will monitor medication adherence using the inhaler's device counter. Visits will be conducted in the Metabolic Bone Diseases Unit. To measure systemic absorption, serum steroid levels will be directly measured.To assess the effects of IGC and dose on the hypothalamic-pituitary-adrenal (HPA) axis, morning (AM) cortisol will be measured at each visit and urinary free cortisol at baseline and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years or at least > 5 years postmenopause (defined as 1 year without a menstrual period)
* No asthma and no history of GC use, either oral or inhaled

Exclusion Criteria:

* Use of oral GCs for > 4 weeks per year in the past 3 years
* History of smoking, to rule out overlapping chronic obstructive pulmonary disease (COPD)
* Other metabolic bone diseases (e.g. hyperparathyroidism, Paget's disease, osteogenesis imperfecta)
* Gastrointestinal Disease (malabsorption, celiac disease, inflammatory bowel disease)
* Endocrinopathies (i.e. untreated thyroid disease, Cushing's syndrome, prolactinoma,)
* Current use of osteoporosis medication (hormone replacement therapy (HRT), raloxifene, bisphosphonates, denosumab)
* Current or past use of teriparatide
* estimated glomerular filtration rate (eGFR)< 45 ml/min calculated by MDRD112 to accommodate mild declines in renal function due to aging
* History of malignancy, except for cured skin cancers
* Diabetes, (HbA1c>6) as this disease is also associated with decreased bone formation
* Osteoporosis by Dual-energy X-ray Absorptiometry (DXA) at any site or an asymptomatic vertebral fracture

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in Osteocalcin | Baseline and 4 weeks
  The primary outcome will be the within-group change in serum osteocalcin from baseline to 4-weeks based on intention-to-treat analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Emily M Stein, MD, Principal Investigator — Columbia University